CLINICAL TRIAL: NCT01613560
Title: Clinical Study of Adjuvant Therapy on Post-menopausal Women With Breast Cancer Under the Guidance of the Results of Preoperative Endocrinotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tao OUYANG (Other)
Responsible Party: Sponsor-Investigator, Tao OUYANG, Chairman of Breast Center, Peking University
Organization: Peking University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCP08
Record Dates: First submitted 2012-05-27; First posted 2012-06-07 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PEPI：2-4 group-A (Experimental)
  Interventions: Drug: AI+chemotherapy adjuvant therapy
- PEPI：2-4 group-B (Active Comparator)
  Interventions: Drug: AI adjuvant therapy
- PEPI：0-1group (Active Comparator)
  Interventions: Drug: AI adjuvant therapy

INTERVENTIONS:
Drug: AI adjuvant therapy — preoperative endocrinotherapy was performed by AI for 4-6 months;surgery;pathological evaluation after surgery;AI adjuvant therapy for 5 years
  Arms: PEPI：0-1group
Drug: AI+chemotherapy adjuvant therapy — preoperative endocrinotherapy was performed by AI for 4-6 months;surgery;pathological evaluation after surgery;AI adjuvant therapy for 5 years after adjuvant chemotherapy
  Arms: PEPI：2-4 group-A
Drug: AI adjuvant therapy — preoperative endocrinotherapy was performed by AI for 4-6 months;surgery;pathological evaluation after surgery;AI adjuvant therapy for 5 years
  Arms: PEPI：2-4 group-B

SUMMARY:
This is a phase II, prospective, multi-center, open-label, non-randomized, controlled study. The objective of this study is to prospectively verify the relation of efficacy of neoadjuvant hormonal therapy, and preliminarily explore the clinical value of complementary adjuvant chemotherapy to predict poor prognosis malignant breast cancer after neoadjuvant endocrinotherapy.

DETAILED DESCRIPTION:
In the decision-making process of a systemic adjuvant therapy for ER-positive/HER2-negative breast cancer, to avoid adjuvant chemotherapy is an attractive but hard choice. On one hand, the result of tamoxifen endocrine therapy combined with adjuvant chemotherapy is superior to tamoxifen endocrine therapy alone for ER-positive breast cancer patients; on the other hand, the benefit that adjuvant chemotherapy provides to breast cancer with high hormone receptor expression is not clear and the tolerance of chemotherapy is much lower than that of endocrinotherapy.

St. Galen consensus on adjuvant therapy for early breast cancer recommends adopting simple endocrinotherapy and avoiding adjuvant chemotherapy for medium- and low- risk breast cancer with hormone receptor highly expressed. However, the results of study P024 and IMPACT suggest that hormone receptor expression is insufficient to predict the effect of endocrinotherapy.

At present, the proven clinical value of neoadjuvant endocrinotherapy is to assist surgery. Consensus recommends neoadjuvant endocrinotherapy for the patients with postmenopausal breast cancer who plan to receive simple adjuvant endocrinotherapy. The current study results show that neoadjuvant endocrinotherapy may be used as an experimental treatment platform, i.e., it can predict the results of adjuvant endocrinotherapy through comprehensive analysis of multiple indexes of the surgery samples after neoadjuvant endocrinotherapy.

By using P024 and IMPACT samples, Ellis et al studied the relation between survival and the test results of surgery samples after neoadjuvant endocrinotherapy, and obtained PEPI (the preoperative endocrine prognostic index). They have preliminarily proved that the PEPI score is relative to RFS (relapse-free survival) of postmenopausal ER-positive breast cancer treated with simple endocrinotherapy and to BCSS (breast cancer-specific survival).

A retrospective study，performed by breast prevention and treatment center in Peking University Cancer Hospital，shows that RFS in PEPI score ≤ 1 group is superior to the PEPI > 1 group after 16 weeks of neoadjuvant endocrinotherapy(p = 0.037), and RFS in effective group (Miller&Payne G1G2G3) is better than that in ineffective group (p=0.001) in terms of pathological evaluation.

The objective of this study is to prospectively verify the relation of efficacy of neoadjuvant hormonal therapy, and preliminarily explore the clinical value of complementary adjuvant chemotherapy to predict poor prognosis malignant breast cancer after neoadjuvant endocrinotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female, not more than 75 years old, judged to have been in menopause by the investigator when enrolled. Refer to the following criteria to determine whether they are postmenopausal breast cancer.

  * Spontaneous amenorrhea for more than 12 months Age ≥ 60 Age < 60, but FSH and E2 reach postmenopausal level.
  * Received bilateral ovariectomy previously
  * Not to define the women using LHRH agonists or antagonists as in postmenopausal state.
* Evidence of primary invasive breast cancer is confirmed by histopathological diagnosis.
* Clinical stage is T2-3N0M0
* ER or PgR are expressed in more than 50 percent of tumour cells, and HER2 is negative.
* No abnormal axillary nodes in ultrasound examination; no evidence of cancer metastasis confirmed by abnormal lymph node puncture pathological examination
* With plan of receiving simple endocrinotherapy and avoiding adjuvant chemotherapy
* No previous breast cancer treatment history
* No other tumors previously; no unstable complications or uncontrolled infection.
* No contraindication for endocrinotherapy with 3rd generation of aromatase inhibitors
* Participate in the trial voluntarily and sign the informed consent form.

Exclusion Criteria:

* Evidence of distant breast cancer metastasis by pathological and imaging diagnosis
* Patients who have a history of other malignant tumors
* With contraindications for 3rd generation of aromatase inhibitors
* Physical condition can not bear the experiment
* Patients who have potential mental, psychological, familial, social, geographic, or other factors that can hinder study regime performance.
* Patients who were treated or are treated with other anti-tumor measures before or during this trial, or planed to participate in other clinical trials.
* Patients who refuse to participate in the trial.

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2012-05-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
RFS | after a follow up of 5 years
  RFS events includes local recurrence, regional recurrence, and distant metastasis resulted from breast cancer
DDFS | after a follow up of 5 years
  DDFS events includes distant metastasis due to breast cancer
BCSS | after a follow up of 5 years
  BCSS events includes death for breast cancer

SECONDARY OUTCOMES:
adverse reaction | during the period of trial (up to 7 years)
  incidence rate of Ⅲ or Ⅳ adverse reaction(according to NCI classification)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ouyang, Doctor, Study Chair — Peking University Cancer Hospital Breast Center
Locations (14):
- China (14):
  - Peking Cancer Hospital & Institute, Beijing, Beijing Municipality
  - 301 Hospital of Pla, Beijing, Beijing Municipality
  - 307 Hospital of Pla, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Cancer Institution and Hospital.Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Wang X, Fan Z, Wang X, He Y, Liu Y, Wang X, Zhang B, Jiang Z, Wang T, Yu Z, Wang F, Liu Y, Li Y, Zhang J, Luo B, Jiang H, Wang T, Xie Y, Li J, Ouyang T. Neoadjuvant endocrine therapy for strongly hormone receptor-positive and HER2-negative early breast cancer: results of a prospective multi-center study. Breast Cancer Res Treat. 2022 Oct;195(3):301-310. doi: 10.1007/s10549-022-06686-1. Epub 2022 Aug 2. PMID 35917052